CLINICAL TRIAL: NCT03982394
Title: Multi-Country Prospective ObserVAtionaL, Cohort Study of Patients With Moderate to Severe Chronic PlaqUE Psoriasis (VALUE)
Brief Title: Observational Study of Patients With Moderate to Severe Chronic Plaque Psoriasis
Acronym: VALUE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P19-377
Record Dates: First submitted 2019-06-10; First posted 2019-06-11 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Chronic Plaque Psoriasis Risankizumab Biologics Psoriasis Vulgaris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants treated with other approved biological therapies: Treatment decision independently made of study enrollment
- Participants treated with Risankizumab: Treatment decision independently made of study enrollment

SUMMARY:
This study will assess the use of risankizumab in adult patients with moderate to severe chronic plaque psoriasis and compare risankizumab to other commonly used biologics.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of moderate to severe chronic plaque-type psoriasis diagnosed by a specialist and presence of moderate to severe psoriasis symptoms according to physician's judgement at time of recruitment.
* Participant starting any approved treatment for psoriasis and physician's decision must be reached prior to recruitment in the study.
* Participant willing to continue with study documentation after cessation of therapy.

Exclusion Criteria:

* Unwillingness or inability to comply with study requirements.
* Participation in an interventional clinical trial, concurrently or within the last 30 days. Participation in a post-market observational study (PMOS) or Registry is acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult subjects with moderate to severe plaque psoriasis.
Sampling Method: Non-Probability Sample
Enrollment: 2759 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who achieved Psoriasis Area and Severity Index (PASI) 90 | From Month 4 to 3 years
  PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination.
Time to first treatment change | From Week 0 (Baseline) to first treatment change
  Identify time to first treatment change including discontinuation, dose escalation and dosing interval shortening

SECONDARY OUTCOMES:
Time to first treatment change rate | At 1 year, 2 year, and 3 year
  Time to first treatment change including discontinuation, dose escalation and dose interval shortening.
Percentage of participants who achieved Static Physicians Global Assessment (sPGA) 0/1 or sPGA 0 | Monthly for up to 3 years
  The sPGA is the physician's current assessment of the average thickness, erythema, and scaling of all psoriatic lesions. sPGA scores demonstrate overall psoriatic disease with a lower score indicating less body coverage. The assessment is considered "static" which refers to the patients disease state at the time of the assessments, without comparison to any of the patient's previous disease states, whether at Baseline or at a previous visit.
Percentage of participants who achieved Psoriasis Area and Severity Index (PASI) 75, 90, or 100 | Monthly for up to 3 years
  PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. Each threshold will be analyzed separately.
Percentage of participants who achieved Absolute PASI<=5, <=3 or <=1 | Monthly for up to 3 years
  Used to assess the benefit of psoriasis therapy. Each threshold will be analyzed separately.
Time to achieve sPGA 0/1 or sPGA 0 | Up to 3 years
  The sPGA is the assessment by the Investigator of the overall disease severity at the time of evaluation. The National Psoriasis Foundation Psoriasis Score version of a static PGA is calculated by averaging the total body erythema, induration, and desquamation scores.
Time to achieve PASI 75, 90,or 100 | Up to 3 years
  PASI 75, 90, or 100 defined as at least a 75%/ 90%/ 100% reduction in PASI relative to Week 0 (Baseline). Each threshold will be analyzed separately.
Percentage of participants who achieve sPGA 0/1 or sPGA 0 at 4 Months and maintained the response status at 1 Year, 2 Years and 3 Years without increasing the dose or shortening the dose interval | At 4 months to 1 year, 2 years, and 3 years
  Percentage of participants who achieve sPGA 0/1 or sPGA 0 at 4 Months and maintained the response status at 1 Year, 2 Years and 3 Years without increasing the dose or shortening the dose interval.
Percentage of participants who achieved PASI 90 or PASI 100 at 4 Months and maintained the response status at 1 Year, 2 Years, and 3 Years without changing the indicated dose or dosing interval | At 4 months and 1 year, 2 years, and 3 years
  Percentage of participants who achieved PASI 90 or PASI 100 demonstrating a 90 or 100% reduction in PASI at 4 Months and maintained the response status at 1 Year, 2 Years, and 3 Years without changing the indicated dose or dosing interval.
Change in PASI | From Week 0 to up to 3 years
  PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination.
Change in Body Surface Area (BSA) | From Week 0 to up to 3 years
  BSA can be used to quantify the severity of psoriasis. A decrease in BSA affected by psoriasis indicates improvement.
Change in Dermatology Quality of Life Index (DLQI) Score | From Week 0 to up to 3 years
  The Dermatology Life Quality Index (DLQI) is the most commonly used quality of life (QoL) assessment tool. The DLQI is a self-administered, ten-question questionnaire used to assess the effect of different skin diseases on a subject's quality of life, overall health, and disability status. Scores range from 0 (not relevant/not at all) to 3 (very much).
Percentage of participants who achieve DLQI 0/1 | Monthly for up to 3 years
  The Dermatology Life Quality Index (DLQI) is the most commonly used quality of life (QoL) assessment tool. The DLQI is a self-administered, ten-question questionnaire used to assess the effect of different skin diseases on a subject's quality of life, overall health, and disability status. The higher the DLQI score, the more quality of life is impaired.
Change in Treatment Satisfaction Questionnaire for Medication (TSQM) score | From Week 0 to up to 3 years
  The Treatment Satisfaction Questionnaire for Medication (TSQM) is a widely used generic measure to assess treatment satisfaction with their medication. This is a 100-point scale with higher scores indicating greater satisfaction with medication and provides scores on four scales - side effects, effectiveness, convenience and global satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (302):
- Argentina (11):
  - Emiliano Baccarini Priv Practice /ID# 218581, Lomas de Zamora, Buenos Aires
  - Hospital Universitario Austral /ID# 217540, Pilar, Buenos Aires
  - Stringa Dermatologia /ID# 218450, Ciudad Autonoma Buenos Aires, Buenos Aires F.D.
  - Private Office Cristina Echeverria /ID# 222082, Ciudad Autonoma Buenos Aires, Buenos Aires F.D.
  - Stat Research /ID# 217185, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Buenos Aires Skin /ID# 217657, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - CEDIC Centro de Investigaciones Clinicas /ID# 217184, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Instituto de Neumonologia y Dermatologia /ID# 217429, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Psoriahue Med Interdisciplinar /ID# 217182, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Professional Skin Care /ID# 218514, Buenos Aires
  - Hospital Italiano /ID# 217000, CABA
- Australia (6):
  - Premier Specialist /ID# 218158, Kogarah, New South Wales
  - Kingsway Dermatology & Aesthetics /ID# 217616, Miranda, New South Wales
  - Northern Dermatology /ID# 218374, Chermside, Queensland
  - Veracity Clinical Research /ID# 217618, Woolloongabba, Queensland
  - Skin Health Institute Inc /ID# 217619, Carlton, Victoria
  - Fremantle Dermatology /ID# 217617, Fremantle, Western Australia
- Austria (9):
  - Medizinische Universitaet Graz /ID# 217702, Graz, Styria
  - Klinikum Wels-Grieskirchen GmbH /ID# 216140, Wels, Upper Austria
  - Klinik Landstrasse /ID# 217684, Vienna, Vienna
  - Medizin am Hauptbahnhof /ID# 218837, Vienna, Vienna
  - EZW HAUT Entzuendungszentrum Wien /ID# 215488, Vienna, Vienna
  - Klinik Hietzing /ID# 217685, Vienna, Vienna
  - Klinik Donaustadt /ID# 218842, Vienna, Vienna
  - Hautarzt Dr. Lukas Kraus /ID# 216139, Dornbirn, Vorarlberg
  - Haut Trattner Dermatologie /ID# 216138, Hainfeld
- Canada (27):
  - Beacon Dermatology Inc /ID# 213524, Calgary, Alberta
  - Duplicate_Stratica Medical /ID# 213526, Edmonton, Alberta
  - Alberta DermaSurgery Centre /ID# 230114, Edmonton, Alberta
  - University of British Columbia - Eye Care Centre, Vancouver General Hospital /ID# 213507, Vancouver, British Columbia
  - SKIN Clinics /ID# 213082, Brandon, Manitoba
  - Winnipeg Clinic /ID# 212134, Winnipeg, Manitoba
  - Dr. Irina Turchin PC Inc. /ID# 212128, Fredericton, New Brunswick
  - Karma Clinical Trials /ID# 213522, St. John's, Newfoundland and Labrador
  - NewLab Clinical Research Inc. /ID# 213521, St. John's, Newfoundland and Labrador
  - Dr. Brown-Maher PMC INC. /ID# 212136, St. John's, Newfoundland and Labrador
  - CCA Medical Research /ID# 214446, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Center /ID# 213081, Barrie, Ontario
  - LEADER Research /ID# 249701, Hamilton, Ontario
  - Lima's Excellence in Allergy and Dermatology Research Inc /ID# 231973, Hamilton, Ontario
  - Hamilton Health Sciences Corporation /ID# 214053, Hamilton, Ontario
  - Dermatrials Research /ID# 213523, Hamilton, Ontario
  - Lynderm Research Inc /ID# 212124, Markham, Ontario
  - Al-Mohammedi Medicine Professional Corporation /ID# 215408, Mississauga, Ontario
  - DermEdge - Queensway East /ID# 213525, Mississauga, Ontario
  - Angela Montgomery Medicine Professional Corporation /ID# 213615, Ottawa, Ontario
  - Dr Melinda Gooderham Medicine Professional Corporation /ID# 212133, Peterborough, Ontario
  - Farheen Mussani Medicine Professional Corporation /ID# 213811, Stoney Creek, Ontario
  - North York Research Inc /ID# 213486, Toronto, Ontario
  - Private Practice - Dr. Kim Papp Clinical Research /ID# 212130, Waterloo, Ontario
  - Dr Maksym Breslavets Medicine Professional Corporation /ID# 213338, Whitby, Ontario
  - Clinique D /ID# 212126, Laval, Quebec
  - Centre de Recherche St-Louis /ID# 216325, Québec, Quebec
- Colombia (9):
  - Fundacion hospitalaria San Vicente de Paul /ID# 222680, Medellín, Antioquia
  - Centro de Inmunología y Genética CIGE SAS /ID# 222685, Medellín, Antioquia
  - IPS Universitaria /ID# 241832, Medellín, Antioquia
  - Fundacion Hospital Universidad del Norte /ID# 223428, Soledad, Atlántico
  - Sociedad de Cirugía de Bogotá- Hospital de San José /ID# 222683, Bogota, Cundinamarca
  - Caja de Compensación Familiar Cafam, Sede Centro de Atención En Salud Cafam Flor /ID# 222660, Bogotá, Cundinamarca
  - Centro Dermatológico Federico Lleras Acosta E.S.E /ID# 222686, Bogotá, Cundinamarca
  - Healthy Medical Center S.A.S /ID# 231909, Zipaquirá, Cundinamarca
  - Ciensalud IPS S.A.S /ID# 244608, Barranqulla
- Czechia (6):
  - Fakultní nemocnice Hradec Králové - Sokolská /ID# 222670, Hradec Králové, Hradec Kralove
  - Nemocnice Ceske Budejovice a.s. /ID# 216310, České Budějovice
  - Fakultni nemocnice Olomouc /ID# 215901, Olomouc
  - Fakultni nemocnice Kralovske Vinohrady /ID# 233184, Prague
  - Sanatorium profesora Arenbergera /ID# 215489, Prague
  - Duplicate_Fakultni Nemocnice v Motole /ID# 215484, Prague
- France (27):
  - Hopital Saint Joseph /ID# 223149, Marseille, Bouches-du-Rhone
  - CHU de Rennes - PONTCHAILLOU /ID# 218248, Rennes, Brittany Region
  - CHU de CAEN - Hopital de la Cote de Nacre /ID# 216245, Caen, Calvados
  - CHU Dijon /ID# 216247, Dijon, Cote-d Or
  - CH Georges Renon /ID# 216174, Niort, Deux-Sevres
  - Hopitaux Drome Nord /ID# 222586, Romans-sur-Isère, Drome
  - CH Valence /ID# 225877, Valence, Drome
  - Hopital de la Cavale Blanche /ID# 216495, Brest, Finistere
  - CH Bigorre - Site de la Gespe /ID# 218563, Tarbes, Hautes-Pyrenees
  - CHU Grenoble - Hopital Michallon /ID# 218437, La Tronche, Isere
  - Ch Chalons En Champagne /Id# 216668, Châlons-en-Champagne, Marne
  - CHR Metz-Thionville - Hopital Bel-Air /ID# 225691, Thionville, Moselle
  - Centre Hospitalier Universitaire de Saint Etienne - Hopital Nord /ID# 216663, St-Priest-en-Jarez, Pays de la Loire Region
  - Centre Hospitalier du Mans /ID# 225729, Le Mans, Sarthe
  - Centre Hospitalier Métropole Savoie - Site Hôpital de Chambéry /ID# 217572, Chambéry, Savoie
  - CHU Amiens-Picardie Site Sud /ID# 216170, Amiens, Somme
  - CH Pontoise - Hopital René Dubos /ID# 216169, Pontoise, Val-d Oise
  - Hôpital d'Instruction des Armées Sainte-Anne /ID# 218888, Toulon, Var
  - Ch Auxerre /Id# 216175, Auxerre, Yonne
  - CH du Pays d'AIX /ID# 216440, Aix-en-Provence
  - Chu Angers /Id# 216244, Angers
  - Hopital Ambroise Pare /ID# 216439, Boulogne-Billancourt
  - Cabinet Dermatologie et Esthetique /ID# 229132, Cannes
  - CH William Morey /ID# 225441, Chalon-sur-Saône
  - CH Annecy Genevois - Site Annecy /ID# 225786, Epagny Metz Tessy
  - C.H. de Bretagne Sud /ID# 216243, Lorient
  - Hôpital d'instruction des armées Bégin /ID# 216167, Saint-Mandé
- Germany (76):
  - Hautarztpraxis Langenau /ID# 213651, Langenau, Baden-Wurttemberg
  - Universitatsklinikum Mannheim /ID# 214569, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 213669, Erlangen, Bavaria
  - Kurzen, Freising, DE /ID# 214567, Freising, Bavaria
  - Beldio Research GmbH /ID# 213958, Memmingen, Bavaria
  - Voelkel, Nuremberg, DE /ID# 213671, Nuremberg, Bavaria
  - Gross/Braeu, Giessen, DE /ID# 213367, Giessen, Hesse
  - Studienzentrum an der Hase GbR Dr. Weyergraf/Dr. Frick/Thomas Heiber /ID# 214466, Bramsche, Lower Saxony
  - Praxis Dres. Kaspari /Schenck /ID# 213649, Hanover, Lower Saxony
  - Breitsprecher, Osnabrueck, DE /ID# 213672, Osnabrück, Lower Saxony
  - Klinikum Rosenhoehe /ID# 215520, Bielefeld, North Rhine-Westphalia
  - Kramer/Mortazawi, Remscheid /ID# 213477, Remscheid, North Rhine-Westphalia
  - Karl, Soest, DE /ID# 214547, Soest, North Rhine-Westphalia
  - Bell, Andernach, DE /ID# 214545, Andernach, Rhineland-Palatinate
  - Grossmann, Koblenz, DE /ID# 214245, Koblenz, Rhineland-Palatinate
  - Universitaetsmedizin Mainz /ID# 222025, Mainz, Rhineland-Palatinate
  - Zentrum fur Hautgesundheit /ID# 222001, Neuwied, Rhineland-Palatinate
  - CMS3 Company for Medical Study /ID# 213676, Selters, Rhineland-Palatinate
  - HMS GmbH Zimmer /ID# 225219, Merzig, Saarland
  - Neubauer, Leipzig, DE /ID# 214548, Leipzig, Saxony
  - Noack-Wiemers, Leipzig, DE /ID# 213654, Leipzig, Saxony
  - Bruecher, Magdeburg, DE /ID# 213476, Magdeburg, Saxony-Anhalt
  - Praxis Dr. Raschke /ID# 225213, Magdeburg, Saxony-Anhalt
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 213670, Kiel, Schleswig-Holstein
  - DermaKiel Allergie und Haut Centrum /ID# 213977, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Jena /ID# 214259, Jena, Thuringia
  - Praxis Dr. Mihaescu /ID# 213483, Augsburg
  - Mauer, Bad Kreuznach, DE /ID# 224876, Bad Kreuznach
  - Hautmedizin Bad Soden /ID# 213956, Bad Soden am Taunus
  - Timmel/Timm/Vorwerk, Bergen /ID# 214552, Bergen
  - Hasert & Hasert, Berlin, DE /ID# 213641, Berlin
  - Hautzentrum Friedrichshain /ID# 213981, Berlin
  - Weihe/Stavermann, Berlin, DE /ID# 214550, Berlin
  - Praxis Dr. med. Alexander Zich /ID# 245751, Berlin
  - Hautarztzentrum Tegel /ID# 214849, Berlin
  - Praxis fuer Innere Medizin/Rheumatologie /ID# 213653, Blaubeuren Abbey
  - Praxis T. Schadeck /ID# 213957, Bogen
  - Barth, Borna, DE /ID# 213643, Borna
  - Schwichtenberg, Bremen, DE /ID# 213650, Bremen
  - Elbe Klinikum Buxtehude /ID# 213366, Buxtehude
  - Praxis Herbst /ID# 222024, Darmstadt
  - Praxis Dr. Sbornik /ID# 213668, Deggendorf
  - Heidlas, Dessau-Rosslau, DE /ID# 217691, Dessau
  - Richter-Huhn, Dresden, DE /ID# 213659, Dresden
  - Praxis Dr. Korge /ID# 213475, Düren
  - Dres. Cesko u. Körber /ID# 214850, Essen
  - Gemeinschaftspraxis Rietkoetter und Jablonka /ID# 213482, Gelsenkirchen
  - Praxis Dr. Lange /ID# 213984, Gera
  - Loth, Gernsbach, DE /ID# 214848, Gernsbach
  - Hautarztpraxis Dr. Viehmann /ID# 213675, Giessen
  - Brinkmann & Partner, Gladbeck, /ID# 214247, Gladbeck
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 222464, Hamburg
  - Dermatologikum Hamburg /ID# 213978, Hamburg
  - Goldbek Medical /ID# 214570, Hamburg
  - Hautarztpraxis Haßberge /ID# 213644, Haßfurt
  - Gemeinschaftspraxis Dres. Anika Hünermund/Mario Pawlak /ID# 213113, Heilbad Heiligenstadt
  - Reinecke, Holzminden, DE /ID# 215081, Holzminden
  - Derma Sana /ID# 214544, Karlsruhe
  - Praxis Dres. Bornemann/Reinerth /ID# 213368, Krefeld
  - Dres. Jacobs & Kollegen /ID# 213652, Kulmbach
  - Hagemeier, Loehne, DE /ID# 214845, Löhne
  - Dlugosz-Wolf, Luedenscheid, DE /ID# 222000, Lüdenscheid
  - Universitaetsklinikum Magdeburg /ID# 215080, Magdeburg
  - Dermatologie Quist-BAG Dres. med. Quist PartG /ID# 214249, Mainz
  - ZENTderma /ID# 213959, Mönchengladbach
  - Duplicate_Praxis Dres. Kloss/Peterburgskiy /ID# 213960, Neuwied
  - Praxis Dr. Konstantin Ertner /ID# 213640, Nuremberg
  - Praxis Dr. Fränken /ID# 214546, Schwelm
  - Praxis Dr. Langhoff /ID# 214253, Schwerin
  - Praxis Dres. Ziegler & Partner /ID# 213647, Stuttgart
  - Braun, Ueberlingen, DE /ID# 213646, Überlingen
  - Barnikol, Waltershausen, DE /ID# 213219, Waltershausen
  - Pfennig, Werdau, DE /ID# 213657, Werdau
  - Moeller, Wiesbaden, DE /ID# 213955, Wiesbaden
  - Hautarztpraxis Dr. med. Matthias Hoffmann /ID# 213444, Witten
  - Franz, Wolfenbuettel, DE /ID# 215355, Wolfenbüttel
- Hungary (4):
  - Pecsi Tudomanyegyetem Klinikai Kozpont /ID# 212960, Pécs, Baranya
  - Debreceni Egyetem-Klinikai Kozpont /ID# 212959, Debrecen, Hajdú-Bihar
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz /ID# 212961, Szombathely, Vas County
  - Szegedi Tudomanyegyetem /ID# 212958, Szeged
- Ireland (3):
  - Tallaght University Hospital /ID# 212999, Tallaght, Dublin, Dublin
  - South Infirmary Victoria University Hospital /ID# 213001, Cork
  - University Hospital Limerick /ID# 216997, Limerick
- Italy (20):
  - Azienda Ospedaliera Universitaria Mater Domini- Campus Salvatore Venuta /ID# 218902, Germaneto, Catanzaro
  - Università degli Studi di Firenze /ID# 221383, Florence, Firenze
  - Ospedale San Martino /ID# 218844, Genoa, Genova
  - ASL 1 Abruzzo - Ospedale regionale San Salvatore /ID# 218719, L’Aquila, L Aquila
  - Sapienza University of Rome - Polo Pontino /ID# 218557, Terracina, Latina
  - IRCCS Istituto Clinico Humanitas /ID# 218560, Rozzano, Lombardy
  - Azienda Ospedaliera Universitaria Federico II /ID# 218808, Naples, Napoli
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli /ID# 218546, Naples, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 219031, Rome, Roma
  - Presidio Columbus-Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Un /ID# 218718, Rome, Roma
  - Azienda Ospedaliero Universitaria delle Marche /ID# 218720, Ancona
  - A.O.U. Consorziale Policlinico di Bari /ID# 218558, Bari
  - ASST degli Spedali Civili di Brescia /ID# 218717, Brescia
  - AOU Policlinico G. Rodolico - San Marco /ID# 219032, Catania
  - IRCCS Policlinico San Donato /ID# 222002, Milan
  - IRCCS Istituto Ortopedico Galeazzi /ID# 218867, Milan
  - Azienda Ospedale-Universita Padova /ID# 221299, Padua
  - Azienda Ospedaliera di Perugia - Ospedale S. Maria della Misericordia /ID# 219033, Perugia
  - Azienda Ospedaliero Universitaria Pisana /ID# 218555, Pisa
  - Azienda ULSS 8 Berica /ID# 218845, Vicenza
- Japan (27):
  - Chukyo Hospital /ID# 213405, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 213363, Nagoya, Aichi-ken
  - Duplicate_Fujita Health University Hospital /ID# 224742, Toyoake-shi, Aichi-ken
  - Matsuyama Red Cross Hospital /ID# 224745, Matsuyama, Ehime
  - Fukuoka University Hospital /ID# 213395, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 215034, Kurume-shi, Fukuoka
  - Asahikawa Medical University Hospital /ID# 213409, Asahikawa-shi, Hokkaido
  - Takagi Dermatological Clinic /ID# 213407, Obihiro-Shi, Hokkaido
  - JR Sapporo Hospital /ID# 213406, Sapporo, Hokkaido
  - Takamatsu Red Cross Hospital /ID# 222875, Takamatsu, Kagawa-ken
  - Takamatsu Red Cross Hospital /ID# 241120, Takamatsu, Kagawa-ken
  - Imamura General Hospital /ID# 228450, Kagoshima, Kagoshima-ken
  - University Hospital Kyoto Prefectural University of Medicine /ID# 213396, Kyoto, Kyoto
  - Kyoto University Hospital /ID# 213404, Kyoto, Kyoto
  - Mie University Hospital /ID# 213387, Tsu, Mie-ken
  - Shinshu University Hospital /ID# 213408, Matsumoto-shi, Nagano
  - University of the Ryukyus Hospital /ID# 213394, Ginowan-shi, Okinawa
  - Kansai Medical University Hospital /ID# 213388, Hirakata-shi, Osaka
  - Shizuoka General Hospital /ID# 224744, Shizuoka, Shizuoka
  - Jichi Medical University Hospital /ID# 213403, Shimotsuke-shi, Tochigi
  - Nippon Medical School Hospital /ID# 213391, Bunkyo-ku, Tokyo
  - St. Lukes International Hospital /ID# 213392, Chuo-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 217125, Shinjuku-ku, Tokyo
  - Japan Community Health care Organization Tokyo Yamate Medical Center /ID# 213389, Shinjuku-ku, Tokyo
  - Nippon Life Saiseikai Public Interest Foundation Nippon Life Hospital /ID# 224743, Osaka
  - The Jikei University School of Medicine /ID# 213393, Tokyo
  - Teikyo University Hospital /ID# 213362, Tokyo
- Mexico (8):
  - Dermatologica Sc /Id# 225449, Tijuana, Estado de Baja California
  - Centro Dermatologico Del Country S de Rl de Cv /Id# 225460, Guadalajara, Jalisco
  - Grupo Clinico Catei Sociedad Civil /Id# 216978, Guadalajara, Jalisco
  - RM Pharma Specialists S.A de C.V. /ID# 225458, Mexico City, Mexico City
  - Consultorio Privado /Id# 225457, Mexico City, Mexico City
  - Clinica Los Arcos Iztapalapa /Id# 216982, Mexico City, Mexico City
  - Centro Especializado en Diabetes, Obesidad y Prevención Cardiovascular (Cedopec) /ID# 216979, Mexico City, Mexico City
  - Neki Servicios Medicos Profesionales S D Rl de Cv /Id# 216977, Toluca
- Netherlands (4):
  - Radboud Universitair Medisch Centrum /ID# 213592, Nijmegen, Gelderland
  - Laurentius Ziekenhuis /ID# 230503, Roermond, Limburg
  - Medisch Centrum Leeuwarden /ID# 215779, Leeuwarden, Provincie Friesland
  - Haaglanden Medisch Centrum /ID# 232063, The Hague
- Poland (4):
  - Panstwowy Instytut Medyczny MSWiA w Warszawie /ID# 225415, Warsaw, Masovian Voivodeship
  - KSW nr1 w Rzeszowie /ID# 225444, Rzeszów, Podkarpackie Voivodeship
  - COPERNICUS Podmiot Leczniczy Sp. z o.o. - Szpital sw. Wojciecha Adalberta /ID# 225446, Gdansk, Pomeranian Voivodeship
  - Labderm S.C. Beata Bergler-Czop, Barbara Sido-Bergler /Id# 225447, Ożarowice, Silesian Voivodeship
- Romania (4):
  - Spitalul Clinic Colentina /ID# 214307, Bucharest
  - Spitalul Clinic Colentina /ID# 224810, Bucharest
  - Spitalul Clinic Colentina /ID# 224811, Bucharest
  - Spitalul Clinic Județean de Urgențe "Sfântul Spiridon" /ID# 214335, Iași
- Saudi Arabia (4):
  - King Abdulaziz Medical City- National Guard Hospital /ID# 224354, Riyadh, Riyadh Region
  - Heraa General Hospital /ID# 217214, Mecca
  - King Saud University Med City /ID# 219065, Riyadh
  - Security Forces Hospital /ID# 221073, Riyadh
- Spain (27):
  - Complejo Hospitalario Universitario de Santiago (CHUS) /ID# 225076, Santiago de Compostela, A Coruna
  - Hospital de Manacor /ID# 225083, Manacor, Balearic Islands
  - Hospital Universitari Son Espases /ID# 233286, Palma de Mallorca, Balearic Islands
  - Hospital Universitario de Puerto Real /ID# 225103, Puerto Real, Cadiz
  - Hospital Universitario Principe de Asturias /ID# 225085, Alcalá de Henares, Madrid
  - Hospital Universitario del Sureste /ID# 226561, Arganda, Madrid
  - Hospital Universitario de Getafe /ID# 225086, Getafe, Madrid
  - Hospital Universitario Severo Ochoa /ID# 225087, Leganés, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 225084, Majadahonda, Madrid
  - Hospital General de Mostoles /ID# 225088, Móstoles, Madrid
  - Hospital Santa María del Rosell /ID# 225100, Cartagena, Murcia
  - Hospital Alvaro Cunqueiro CHUVI /ID# 225077, Vigo, Pontevedra
  - Hospital Universitario de Bajadoz /ID# 225091, Badajoz
  - Hospital Universitario Virgen de las Nieves /ID# 225107, Granada
  - Hospital Juan Ramon Jimenez /ID# 225105, Huelva
  - Hospital de Leon /ID# 226559, León
  - Hospital Universitario Lucus Augusti /ID# 233282, Lugo
  - Hospital General Universitario Gregorio Maranon /ID# 231664, Madrid
  - Hospital Universitario Ramon y Cajal /ID# 225093, Madrid
  - Hospital Universitario 12 de Octubre /ID# 238474, Madrid
  - Hospital San Telmo /ID# 233283, Palencia
  - Hospital Universitario de Salamanca /ID# 225078, Salamanca
  - Hospital Universitario Virgen de Valme /ID# 225104, Seville
  - Hospital Virgen de la Concha /ID# 233285, Zamora
  - Hospital Clinico Universitario Lozano Blesa /ID# 231663, Zaragoza
  - Hospital Universitario Miguel Servet /ID# 225080, Zaragoza
  - Hospital Royo Villanova /ID# 231665, Zaragoza
- Switzerland (5):
  - University Hospital Basel /ID# 212744, Basel Town, Canton of Basel-City
  - Waldhotel Health & Medical Excellence /Id# 212743, Obbürgen, Canton of Nidwalden
  - Haut. Venen. Allergie. Zentrum Brunnehof /ID# 212742, Uster, Canton of Zurich
  - University Hospital Zurich /ID# 216539, Zurich, Canton of Zurich
  - Inselspital, Universitaetsspital Bern /ID# 212741, Bern
- United Arab Emirates (5):
  - Mediclinic Khalifa Branch /ID# 217871, Abu Dhabi
  - New Medical Center Hospital /ID# 223681, Abu Dhabi
  - Skmc /Id# 217873, Abu Dhabi
  - Tawam Hospital /ID# 217872, Abu Dhabi
  - Mediclinic Welcare Hospital /ID# 223683, Dubai
- United Kingdom (16):
  - Addenbrookes Hospital /ID# 215972, Cambridge, Cambridgeshire
  - Western General Hospital - NHS Lothian /ID# 249287, Edinburgh, Edinburgh, City of
  - Hammersmith Hospital /ID# 215978, London, England
  - The Queen Elizabeth Hospital, Kings Lynn NHS Foundation Trust /ID# 215476, Kings Lynn, Norfolk
  - York Hospital /ID# 227940, York, North Yorkshire
  - Northampton General Hospital NHS Trust /ID# 249297, Northampton, Northamptonshire
  - West Suffolk Hospital /ID# 249283, Bury St Edmunds, Suffolk
  - Frimley Health NHS Foundation Trust /ID# 215976, Camberley, Surrey
  - Kingston Hospital NHS Foundation Trust /ID# 215973, Kingston upon Thames, Surrey
  - Kingston Hospital NHS Foundation Trust /ID# 230856, Kingston upon Thames, Surrey
  - Cwm Taf Morgannwg University Health Board /ID# 215974, Bridgend, Wales
  - Ulster Hospital - South Eastern Health & Social Care Trust /ID# 215477, Belfast
  - The Dudley Group NHS Foundation Trust /ID# 215839, Dudley
  - Sandwell and West Birmingham Hospitals NHS Trust /ID# 249294, Lyndon
  - Northern Care Alliance NHS Group /ID# 218589, Manchester
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 215479, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thaci D, Ohtsuki M, Maul JT, Szegedi A, Luna PC, Lynde CW, Soliman AM, Wang H, Kaufmann C, Ashley DG, Madihlaba T, Rubant S, Papp KA. Real-World Effectiveness of Risankizumab in Patients with Moderate-to-Severe Psoriasis: Interim Analysis from the VALUE Global Prospective Post-marketing Observational Study at 25 Months. Dermatol Ther (Heidelb). 2025 Feb;15(2):381-394. doi: 10.1007/s13555-025-01342-0. Epub 2025 Feb 4. PMID 39904971
- See also: Related info — https://www.rxabbvie.com/